CLINICAL TRIAL: NCT05095428
Title: The PARTS Study: A Pilot Randomized Controlled Trial of the PARTS Intensive IFS Program vs. a Nature-based Stress Reduction Program for PTSD in a Community Mental Health Clinic
Brief Title: Program for Alleviating and Resolving Trauma and Stress 2
Acronym: PARTS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Foundation for Self Leadership (Other)
Responsible Party: Principal Investigator, Zev Schuman Olivier, Director, Center for Mindfulness and Compassion and Director of Addiction Research, Cambridge Health Alliance
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHA-IRB-21-22-18
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; stress; RCT
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be unaware of study hypotheses or arms and will be told the study is for stress reduction among people with trauma/PTSD.
  The staff member responsible for final determination of study eligibility will be blinded to the randomization sequence.
  The Data Analyst and methodologist will be blinded to participant identity prior to and during randomization and analysis.
  The PI will be blinded to participant randomization status for the duration of the study.
  Medical Review Officer: The MRO will not be blinded and will be responsible for advising on adverse events.
  Independent Evaluators conducting the CAPS-5 assessments will be blinded to the participants' randomization status. To protect this, independent CAPS-5 evaluators will be located separately from group leaders and therapists. In the event of an unintentional unblinding, a new rater will be assigned to assess the relevant participant(s).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARTS (Experimental): The Program for Alleviating and Resolving Trauma and Stress (PARTS) Program is a 16-week group intervention model of Internal Family Systems (IFS), with 8 individual IFS clinical sessions on a biweekly basis, developed to resolve and alleviate trauma and stress for individuals diagnosed with PTSD.
  Interventions: Behavioral: PARTS Program
- NBSR-T (Active Comparator): The Nature Based Stress Reduction for Trauma Survivors (NBSR-T) Program is a 16-week nature-based group intervention model, with 8 individual non-IFS clinical sessions on a biweekly basis, developed as an attention placebo control for individuals diagnosed with PTSD.
  Interventions: Behavioral: NBSR-T Program

INTERVENTIONS:
Behavioral: PARTS Program — The PARTS Program is a 16-week group intervention model of Internal Family Systems (IFS), with 8 individual IFS clinical sessions on a biweekly basis, developed to resolve and alleviate trauma and stress for individuals diagnosed with PTSD.
  Arms: PARTS
Behavioral: NBSR-T Program — The NBSR-T Program is a 16-week nature-based group intervention model, with 8 individual non-IFS clinical sessions on a biweekly basis, developed as an attention placebo control for individuals diagnosed with PTSD.
  Arms: NBSR-T

SUMMARY:
This pilot RCT will test the preliminary efficacy of an intensive group model of Internal Family Systems (IFS) called the Program for Alleviating and Resolving Trauma and Stress (PARTS) compared with a Nature-Based Stress Reduction for Trauma Survivors (NBSR-T) attention placebo control group at reducing PTSD symptom severity measured by Clinician-Administered PTSD Scale (CAPS-5). In addition, the effects of the interventions on self-reported PTSD symptoms, disassociation, and disturbances of self-organization (DSO), as well as mechanisms of emotion regulation, decentering and self-compassion will be secondary outcomes.

DETAILED DESCRIPTION:
The investigators will conduct a pilot RCT to test the preliminary efficacy of the Program for Alleviating and Resolving Trauma and Stress (PARTS) compared with a Nature-Based Stress Reduction for Trauma Survivors (NBSR-T) control group at reducing PTSD symptom severity measured by Clinician-Administered PTSD Scale (CAPS-5).

Secondary clinical outcomes include the effects of the intervention on self-reported PTSD symptoms (PCL-5; CAT-PTSD), disassociation (MDI), and disturbances of self-organization (ITQ). Secondary mechanistic outcomes include emotion regulation (DERS), self-compassion (SCS-SF), and decentering (EQ-D) .

Exploratory aims of the study are to investigate the effects on depression (CAT-DI), mental health (CAT-MH scales), self-trauma fusion (PRISM-D), perceived stress (PSS), internalized stigma (ISMI), and interoception (MAIA-2). Additional exploratory outcomes include changes in outcome variables among PTSD subjects with baseline DSO and those without DSO as defined by the International Trauma Questionnaire (ITQ).

ELIGIBILITY:
Inclusion Criteria:

* Be able to bill insurance for individual psychotherapy at CHA;
* Be a current patient of CHA primary care, behavioral health care or CHA MINDWell;
* Have a current diagnosis of PTSD OR a CAT-MH PTSD score >58;
* Have sufficient English fluency and literacy skills to understand the consent process, procedures and questionnaires and have the ability to provide written informed consent;
* Have access to the internet and an electronic device with adequate data capacity; to complete questionnaires online and attend online videoconference groups;
* Must be available and willing to attend the scheduled online group sessions for 16 weeks; and must be available and willing to complete the online computerized assessments and phone interviews.

Exclusion Criteria:

* Inability to complete an informed consent assessment AND/OR inability to complete baseline study assessment procedures (due to cognitive deficit, non-proficiency in English literacy, or any other reason);
* Current participation in another experimental research study;
* Expected medical hospitalization in six months from the date of enrollment;
* Expected incarceration in six months from the date of enrollment;
* Individuals who are pregnant with a due date within 26 weeks after study consent;
* Insufficient level of severity of PTSD symptoms: CAPS-5 SEV2 Total score less than 26; PTSD score of less than 31 on the PTSD Checklist for DSM-V (PCL-5)8 at screening visit;
* Inability to participate safely in the study intervention and without disrupting the group (in the opinion of principal investigator OR meeting any of the following criteria):
* Past year history of a psychotic disorder or clinician confirmed active psychosis (Severe level of psychosis on PSY-S-CAT > 30 will trigger the requirement of a clinical assessment prior to participation in the program)
* Bipolar I disorder history or severe level of mania on CAT-MH5 (>70)
* Acute suicidality or self-injurious behavior
* Severe depression, indicated by CAT-DI > 755,65
* Acute homicidality with plan and/or intent;
* Hospitalization for suicide attempt or self-harm within three months of the enrollment period;
* Severe Borderline Personality Disorder or other severe personality disorder that may lead to disruptions within the group; and/or
* Moderate or severe Substance Use Disorder. In addition, use of or positive toxicology for illicit drugs (e.g., cocaine, opioids, etc.) or non-prescribed controlled medications (i.e., opioids, stimulants, or benzodiazepines) in the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline CAPS-5 at 16 Weeks | Week 16
  The primary aim of this study is to examine the preliminary efficacy of a live-online version of the PARTS program on PTSD symptoms measured by reduction in CAPS-5 over 16 weeks. The CAPS-5 is a 30-item questionnaire administered by a trained interviewer and is considered the "gold standard" assessment for PTSD diagnosis and symptoms as defined by the DSM-5. This measure also assesses the duration of symptoms, impact of symptoms on aspects of the participant's life, and if the participant meets criteria for the dissociative subtype of PTSD.

SECONDARY OUTCOMES:
Change from Baseline Self-reported PTSD symptoms (PCL-5) at 16 Weeks | Week 16
  Participants will be sent a link to complete the PTSD Checklist for DSM-5 (PCL-5), which is a self-report measure with 20 items, which is designed to measure PTSD symptom severity over the past month as measured by the DSM-5, in combination with additional diagnostic tools.
Change from Baseline Self-reported PTSD symptoms (CAT-PTSD) at 16 Weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome refers to the CAT-PTSD severity score.
Change from Baseline Disturbances of Self Organization -- International Trauma Questionnaire (ITQ-DSO-9) at 16 Weeks | Week 16
  The International Trauma Questionnaire (ITQ) is the first instrument designed to capture the ICD-11 PTSD and Complex PTSD (CPTSD) diagnoses. The last 6 items measure DSO symptoms characteristic of ICD-11 CPTSD. Each set of items have 3 severity of impact on functioning questions. The ITQ-DSO-9 includes just the 6 DSO items with 3 severity questions. The ITQ-DSO-9 will be used monthly for self-report of changes in DSO symptoms.
Change from Baseline Difficulties in Emotion Regulation (DERS) Scale at 16 Weeks | Week 16
  The DERS is a 36-item self-report scale designed to assess emotional dysregulation. The scale assess 6 aspects of emotional dysregulation: non-acceptance of emotional responses ("When I'm upset, I become embarrassed for feeling that way"), difficulties engaging in goal directed behavior ("When I'm upset, I have difficulty thinking about anything else"), impulse control difficulties ("When I'm upset, I lose control over my behaviors"), lack of emotional awareness ("When I'm upset, I take time to figure out what I'm really feeling (reverse-scored)", limited access to emotion regulation strategies ("When I'm upset, it takes me a long time to feel better"), and lack of emotional clarity ("I have no idea how I am feeling").
Change from Baseline Multiscale Dissociation Inventory (MDI) at 16 Weeks | Week 16
  The MDI is a 30-item self-report inventory measuring frequency of dissociative symptoms (e.g., depersonalization, derealization, emotional constriction, identity dissociation, etc.)
Change from Baseline Self-Compassion Scale (SCS-SF) at 16 Weeks | Week 16
  The SCS-SF is an abbreviated 12-item form of the original 26-item Self-Compassion Scale. This scale evaluates 6 different aspects of self-compassion: Self-Kindness (e.g., ''I try to be understanding and patient toward those aspects of my personality I don't like''), Self-Judgment (e.g., ''I'm disapproving and judgmental about my own flaws and inadequacies''), Common Humanity (e.g., ''I try to see my failings as part of the human condition''), Isolation (e.g., ''When I feel inadequate in some way, I try to remind myself that feelings of inadequacy are shared by most people"), Mindfulness (e.g., ''When something painful happens I try to take a balanced view of the situation''), and Over-Identification (e.g., ''When I'm feeling down I tend to obsess and fixate on everything that's wrong.''). The scale is scored on a 5-point Likert scale (1 = Almost never; 5 = Almost always), and negative subscale items are reverse scored.
Change from Baseline Decentering (EQ-D) at 16 weeks | Week 16
  The EQ-D is an 11-item scale representing the Decentering items of the Experiences Questionnaire.

OTHER OUTCOMES:
Change from Baseline Pictorial Representation of Illness and Self Measure Drawaing (PRISM-D) --Trauma at 16 Weeks | Week 16
  drawing version of the PRISM, a virtual visual method to assess the global burden of illness.
Change from Baseline Depression (CAT-DI) at 16 Weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assess depression severity with the CAT-DI.
Change from Baseline Perceived Stress Scale (PSS-4) at 16 Weeks | Week 16
  The PSS-4 uses 4 items to measure the degree to which situations in life are stressful, evaluating how overloaded, unpredictable, and uncontrollable one finds one's life. Each item is scored on a 5-point Likert scale from 0 (Never) to 4 (Very often).
Change from Baseline Multidimensional Assessment of Interoceptive Awareness (MAIA-2) at 16 Weeks | Week 16
  The MAIA-2 is a 37-item self-report scale designed to assess multiple aspects of interoception and interoceptive awareness (e.g., body trusting).
Change from Baseline Internalized Stigma of Mental Illness (ISMI) at 16 weeks | Week 16
  The ISMI is a 29-item measure with five subscales (e.g., alienation, stereotype endorsement, perceived discrimination, etc.)
Change from Baseline CAT-Anx at 16 weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assessed with scales for CAT-Anxiety.
Change from Baseline CAT-Mania/Hypomania at 16 weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assessed with scales for CAT-M/HM.
Change from Baseline CAT-SUD at 16 weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assessed with scales for CAT-SUD.
Change from Baseline CAT-Psychosis at 16 weeks | Week 16
  Participants will be sent a link to complete the CAT-MH (Computer Adaptive Testing for Mental Health) interview on a computer, tablet or phone. This outcome will assessed with scales for CAT-PSY.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, M.D., Principal Investigator — Center for Mindfulness and Compassion
Locations (1):
- Cambridge Health Alliance Center for Mindfulness and Compassion, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Eisen SV, Schultz MR, Ni P, Haley SM, Smith EG, Spiro A, Osei-Bonsu PE, Nordberg S, Jette AM. Development and Validation of a Computerized-Adaptive Test for PTSD (P-CAT). Psychiatr Serv. 2016 Oct 1;67(10):1116-1123. doi: 10.1176/appi.ps.201500382. Epub 2016 Jun 1. PMID 27247175
- [Background] Briere J, Weathers FW, Runtz M. Is dissociation a multidimensional construct? Data from the Multiscale Dissociation Inventory. J Trauma Stress. 2005 Jun;18(3):221-31. doi: 10.1002/jts.20024. PMID 16281216
- [Background] Achtyes ED, Halstead S, Smart L, Moore T, Frank E, Kupfer DJ, Gibbons R. Validation of Computerized Adaptive Testing in an Outpatient Nonacademic Setting: The VOCATIONS Trial. Psychiatr Serv. 2015 Oct;66(10):1091-6. doi: 10.1176/appi.ps.201400390. Epub 2015 Jun 1. PMID 26030317
- [Background] Raes F, Pommier E, Neff KD, Van Gucht D. Construction and factorial validation of a short form of the Self-Compassion Scale. Clin Psychol Psychother. 2011 May-Jun;18(3):250-5. doi: 10.1002/cpp.702. Epub 2010 Jun 8. PMID 21584907
- [Background] Mitchell AM, Crane PA, Kim Y. Perceived stress in survivors of suicide: psychometric properties of the Perceived Stress Scale. Res Nurs Health. 2008 Dec;31(6):576-85. doi: 10.1002/nur.20284. PMID 18449942
- [Background] Mehling WE, Acree M, Stewart A, Silas J, Jones A. The Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-2). PLoS One. 2018 Dec 4;13(12):e0208034. doi: 10.1371/journal.pone.0208034. eCollection 2018. PMID 30513087
- [Background] Gratz, K.L., Roemer, L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26, 41-54 (2004). https://doi.org/10.1023/B:JOBA.0000007455.08539.94
- [Background] Kok T, De Haan HA, Sensky T, van der Meer M, De Jong CAJ. Using the Pictorial Representation of Illness and Self Measure (PRISM) to Quantify and Compare Suffering From Trauma and Addiction. J Dual Diagn. 2017 Apr-Jun;13(2):101-108. doi: 10.1080/15504263.2017.1293867. Epub 2017 Feb 22. PMID 28368709
- [Background] Buchi S, Villiger P, Kauer Y, Klaghofer R, Sensky T, Stoll T. PRISM (Pictorial Representation of Illness and Self Measure)- a novel visual method to assess the global burden of illness in patients with systemic lupus erythematosus. Lupus. 2000;9(5):368-73. doi: 10.1191/096120300678828479. PMID 10878730
- [Derived] Joss D, Comeau A, Chevannes R, Parry G, Rea HS, Barria J, Bumpus C, Rector A, Rajan A, Rosansky J, Rice FK, Ward MC, Tobiasz Veltz L, Ally D, Rosenberg LG, Sweezy M, Lovas D, Schuman-Olivier Z. A randomized controlled trial of an online group-based internal family systems treatment for posttraumatic stress disorder: The Program for Alleviating and Resolving Trauma and Stress (PARTS) study. Psychol Trauma. 2026 Jan 29. doi: 10.1037/tra0002089. Online ahead of print. PMID 41609644